CLINICAL TRIAL: NCT00782431
Title: Phase 3 Double Blind Clinical Study of Effectiveness and Safety of Vero Cell-Derived, Trivalent, Seasonal Influenza Vaccine in Adults Aged 50 Years and Older
Brief Title: Immunogenicity and Safety Study of an Inactivated Influenza Vaccine (Split Virus, Vero Cell Derived) in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 720801
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vero cell-derived, trivalent, seasonal influenza vaccine
  Interventions: Biological: Vero cell derived, trivalent, seasonal influenza vaccine
- 2 (Active Comparator): Licensed egg-derived, trivalent seasonal influenza vaccine
  Interventions: Biological: Licensed egg-derived, trivalent seasonal influenza vaccine

INTERVENTIONS:
Biological: Vero cell derived, trivalent, seasonal influenza vaccine — Single intramuscular injection
  Arms: 1
Biological: Licensed egg-derived, trivalent seasonal influenza vaccine — Single intramuscular injection
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the effectiveness (seroprotection and seroconversion as measured by the hemagglutination inhibition [HI] assay) of an investigational Vero cell-derived, trivalent, seasonal influenza vaccine in adults 50 years of age and older. Subjects will be randomized in a double-blind fashion to receive a single intramuscular injection of either the investigational vaccine or a licensed egg-derived seasonal influenza vaccine. Blood will be drawn from all subjects for a determination of HI antibody titers on Days 0 and 21, body temperature and injection site reactions will be monitored daily for 7 days. In addition, subjects will be monitored for adverse events and rises in body temperature until Day 21 and again until Day 180.

ELIGIBILITY:
Inclusion Criteria:

* Are 50 years of age or older on the day of screening
* Have an understanding of the study, agree to its provisions, have the ability to adhere to the provisions of the study and give written informed consent prior to study entry
* If female and capable of bearing children,have a negative urine pregnancy test result within 24 hours prior to the vaccination on Study Day 0 and agree to employ adequate birth control measures.

Exclusion Criteria:

* History of severe allergic reaction or anaphylaxis to egg protein or any other component of the Vero cell-derived influenza vaccine or the egg-derived influenza vaccine
* Oral temperature of >= 99.5°F (37.5°C) on the day of vaccination in this study (Note: Subjects meeting this exclusion criterion may be rescheduled for vaccination and study entry at a later date if certain requirements [in the study protocol] are met)
* Rash or dermatologic condition or tattoos which may interfere with injection site reaction rating
* Blood transfusion or immunoglobulins received within 90 days of study entry
* Live vaccine received within 4 weeks or inactivated vaccine or subunit vaccine received within 2 weeks of study entry
* Previous vaccination against influenza for the 2008/2009 northern hemisphere influenza season
* Functional or surgical asplenia (e.g. from a history of hemoglobinopathies, leukemias, or lymphomas)
* Diagnosed immunodeficiency as a result of a pathological condition
* Pharmacologically induced immunodeficiency as a result of prescribed administration of corticosteroids (e.g., any systemic administration of corticosteroids or an inhaled dose equivalent to 800 mg of beclomethasone dipropionate) or chemotherapeutics or as a result of radiation therapy or any other modality capable of altering normal immunologic response
* Known or suspected problem with drug or alcohol abuse
* Investigational drug received within 6 weeks prior to study entry or concurrent participating in a clinical study that includes the administration of an investigational product
* Subjects who are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, spouse/partner, siblings, parents) as well as employees of the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3208 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Benchmark Research, San Francisco, Sacramento, California
  - California Research Foundation, San Diego, California
  - Benchmark Research San Francisco, San Francisco, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Heartland Research Associates LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research Inc., Rochester, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Omega Medical Research, Warwick, Rhode Island
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Clinical Research Associates, Inc. - Nashville, Nashville, Tennessee
  - Benchmark Research Austin, Austin, Texas
  - Benchmark Research Ft. Worth, Fort Worth, Texas
  - Research Across America, Plano, Texas
  - Benchmark Research San Angelo, San Angelo, Texas
  - Pi-Coor Clinical Research, Fairfax, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia

REFERENCES:
- [Derived] Ehrlich HJ, Berezuk G, Fritsch S, Aichinger G, Singer J, Portsmouth D, Hart MK, El-Amin W, Kistner O, Barrett PN. Clinical development of a Vero cell culture-derived seasonal influenza vaccine. Vaccine. 2012 Jun 19;30(29):4377-86. doi: 10.1016/j.vaccine.2011.11.114. Epub 2011 Dec 13. PMID 22172502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was divided into Part A and Part B and two age strata, 50-64 and 65 and older. Part A began when the first subject consented to participate in the study and ended when the last subject completed Day 21. Part B began after the first subject completed Day 21 and ended when the last subject completed Day 180. All subjects were randomized to receive a single IM injection of seasonal VCIV or licensed EIV. Only subjects that completed Part A were allowed to enroll in Part B.
Groups:
- VCIV (50-64 Years): Vero cell derived, trivalent, seasonal influenza vaccine (VCIV) on Day 1 Subjects aged 50 to 64 years of age
- VCIV (65+ Years): Vero cell derived, trivalent, seasonal influenza vaccine (VCIV) on Day 1 Subjects aged 65 years of age and older
- EIV (50-64 Years): Licensed egg derived, trivalent seasonal influenza vaccine (EIV) on Day 1 Subjects aged 50 to 64 years of age
- EIV (65+ Years): Licensed egg derived, trivalent seasonal influenza vaccine (EIV) on Day 1 Subjects aged 65 years of age and older
- VCIV + EIV (50-64 Years): Subjects administered VCIV on Day 1 and accepted offer to be vaccinated received EIV after Day 21 at a time convenient to the subject.
  Subjects aged 50 to 64 years of age
- VCIV + EIV (65+ Years): Subjects administered VCIV on Day 1 and accepted offer to be vaccinated received EIV after Day 21 at a time convenient to the subject.
  Subjects aged 65 years of age and older
Period: Part A
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years) | VCIV + EIV (50-64 Years) | VCIV + EIV (65+ Years)
Started | 839 | 478 | 229 | 137 | 923 | 602
Completed | 829 | 474 | 227 | 136 | 923 | 602
Not Completed | 10 | 4 | 2 | 1 | 0 | 0
Period: Part B
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years) | VCIV + EIV (50-64 Years) | VCIV + EIV (65+ Years)
Started | 828 | 474 | 227 | 136 | 923 | 602
Completed | 804 | 458 | 227 | 134 | 916 | 600
Not Completed | 24 | 16 | 0 | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Population: Study was divided into Part A and Part B and two age strata, 50-64 and 65 and older. Part A began when the first subject consented to participate in the study and ended when the last subject completed Day 21. All subjects were randomized to receive a single IM injection of seasonal VCIV or licensed EIV. Only subjects that completed Part A were allowed to enroll in Part B. Per SAP, all analysis are performed by treatment group and age stratum.
Groups:
- VCIV (50-64 Years): Vero cell derived, trivalent, seasonal influenza vaccine (VCIV) Subjects aged 50 to 64 years of age
- VCIV (65+ Years): Vero cell derived, trivalent, seasonal influenza vaccine (VCIV) Subjects aged 65 years of age and older
- EIV (50-64 Years): Licensed egg derived, trivalent seasonal influenza vaccine (EIV) Subjects aged 50 to 64 years of age
- EIV (65+ Years): Licensed egg derived, trivalent seasonal influenza vaccine (EIV) Subjects aged 65 years of age and older
- Total: Total of all reporting groups
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years) | Total
Number analyzed (Participants) | 1762 | 1080 | 229 | 137 | 3208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1762 | 0 | 229 | 0 | 1991
  >=65 years | 0 | 1080 | 0 | 137 | 1217
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (4.29) | 71.4 (5.45) | 56.7 (4.56) | 71 (5.87) | 63.8 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1068 | 478 | 91 | 64 | 1701
  Male | 694 | 602 | 138 | 73 | 1507
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 159 | 58 | 15 | 9 | 241
  Not Hispanic or Latino | 1603 | 1022 | 214 | 128 | 2967
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 0 | 1 | 0 | 14
  Asian | 19 | 7 | 5 | 0 | 31
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 0 | 0 | 6
  Black or African American | 217 | 62 | 25 | 6 | 310
  White | 1497 | 1008 | 198 | 131 | 2834
  More than one race | 7 | 1 | 0 | 0 | 8
  Unknown or Not Reported | 4 | 1 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 1762 | 1080 | 229 | 137 | 3208
Weight (kg) [Mean (Standard Deviation); unit: kg] | 85.6 (21.06) | 82.1 (18.53) | 86.4 (21.38) | 81.2 (15.93) | 83.83 (19.31)
Height (cm) [Mean (Standard Deviation); unit: cm] | 168.9 (9.93) | 167.8 (9.71) | 168.8 (9.7) | 167.9 (10.35) | 168.36 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seroconversion Antibody Titer
Description: The rate of subjects vaccinated that demonstrate seroconversion via hemagglutination inhibition (HI) antibody titer to each of the three antigens contained in the vaccine 21 days after vaccination. Seroconversion is defined as a ≥ 4-fold increase in HI antibody titer from baseline or a HI antibody titer ≥ 40 when there is no detectable HI antibody titer (HI antibody titer < 10) at baseline.
Time Frame: 21 days
Population: Intent-to-treat dataset contains all randomized and vaccinated subjects with immunogenicity data available at baseline and Day 21 for at least one strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years)
Number analyzed (Participants) | 1730 | 1066 | 221 | 134
percentage of participants
  A/H1N1 | 47.1 [44.7 to 49.5] | 36.8 [33.9 to 39.7] | 63.8 [57.1 to 70.1] | 37.3 [29.1 to 46.1]
  A/H3N2 | 68.3 [66.1 to 70.5] | 58.1 [55 to 61.1] | 85.1 [79.7 to 89.5] | 67.9 [59.3 to 75.7]
  B | 46.6 [44.2 to 49] | 36.3 [33.4 to 39.3] | 62.9 [56.2 to 69.3] | 51.5 [42.7 to 60.2]

2. Primary Outcome: Percentage of Subjects With Seroprotective Antibody Titer
Description: The rate of subjects vaccinated that achieve a reciprocal HI antibody titer of 40 or higher 21 days after vaccination for each of the three antigens contained in the vaccine.
Time Frame: 21 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years)
Number analyzed (Participants) | 1730 | 1066 | 221 | 134
percentage of participants
  A/H1N1 Day 1 | 29.6 [27.5 to 31.8] | 35.3 [32.4 to 38.2] | 26.7 [21 to 33] | 36.6 [28.4 to 45.3]
  A/H1N1 Day 21 | 74.3 [72.2 to 76.4] | 72.6 [69.8 to 75.3] | 86.9 [81.7 to 91] | 75.4 [67.2 to 82.4]
  A/H3N2 Day 1 | 43.1 [40.8 to 45.5] | 58 [54.9 to 61] | 44.8 [38.1 to 51.6] | 51.5 [42.7 to 60.2]
  A/H3N2 Day 21 | 90 [88.5 to 91.4] | 91.3 [89.4 to 92.9] | 95.9 [92.4 to 98.1] | 95.5 [90.5 to 98.3]
  B Day 1 | 45.7 [43.4 to 48.1] | 49.1 [46 to 52.1] | 42.1 [35.5 to 48.9] | 52.2 [43.4 to 60.9]
  B Day 21 | 86.2 [84.5 to 87.8] | 82.6 [80.2 to 84.9] | 93.7 [89.6 to 96.5] | 94.8 [89.5 to 97.9]

3. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titer for Each of the Three Antigens Contained in the Vaccine at Day 21 After Vaccination
Time Frame: 21 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: HIA Titers
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years)
Number analyzed (Participants) | 1730 | 1066 | 221 | 134
HIA Titers
  A/H1N1 Day 1 | 17.2 [16.3 to 18.2] | 20.3 [18.9 to 21.7] | 15.5 [13.4 to 18] | 20.9 [17.3 to 25.3]
  A/H1N1 Day 21 | 79.5 [74.1 to 85.3] | 67.2 [62 to 72.9] | 106.5 [90.8 to 125] | 68.7 [56.3 to 83.9]
  A/H3N2 Day 1 | 24.7 [23 to 26.4] | 41.6 [38 to 45.5] | 23.8 [19.9 to 28.6] | 39.7 [30.5 to 51.5]
  A/H3N2 Day 21 | 221.2 [205.5 to 238.1] | 234.9 [214.7 to 256.9] | 358.6 [297.2 to 432.8] | 320 [252.6 to 405.5]
  B Day 1 | 28.6 [26.8 to 30.6] | 31.4 [29 to 34] | 24.6 [20.6 to 29.4] | 33.1 [26.8 to 41]
  B Day 21 | 122.5 [115.1 to 130.4] | 95.5 [88.4 to 103.2] | 181.6 [155 to 212.7] | 151.4 [124.9 to 183.6]

4. Secondary Outcome: Change of Hemagglutination Inhibition (HI) Antibody Titer at Day 21 Compared to Baseline
Description: Change in geometric mean of titers at day 21 compared to baseline
Time Frame: 21 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: HIA Titers
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years)
Number analyzed (Participants) | 1730 | 1066 | 221 | 134
HIA Titers
  A/H1N1 | 4.61 [4.31 to 4.94] | 3.32 [3.07 to 3.59] | 6.87 [5.69 to 8.31] | 3.29 [2.7 to 4]
  A/H3N2 | 8.96 [8.33 to 9.64] | 5.65 [5.19 to 6.15] | 15.04 [12.4 to 18.25] | 8.07 [6.21 to 10.48]
  B | 4.28 [4.01 to 4.57] | 3.04 [2.83 to 3.27] | 7.37 [6.09 to 8.93] | 4.57 [3.63 to 5.74]

5. Secondary Outcome: Rate of Subjects Experiencing Any Injection Site Reactions Until the Day 21 Visit After Vaccination
Time Frame: 21 days
Population: Safety dataset contains all vaccinated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years)
Number analyzed (Participants) | 1762 | 1080 | 229 | 137
Participants | 625 | 222 | 73 | 34

6. Secondary Outcome: Rate of Subjects Experiencing Systemic Reactions Until the Day 21 Visit After Vaccination
Time Frame: 21 days
Population: Safety dataset contains all vaccinated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years)
Number analyzed (Participants) | 1762 | 1080 | 229 | 137
Participants | 985 | 465 | 119 | 53

7. Secondary Outcome: Rate of Subjects Experiencing Any Systemic Adverse Events During the Entire 180 Day Follow-up Period
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years) | VCIV + EIV (50-64 Years) | VCIV + EIV (65+ Years)
Number analyzed (Participants) | 828 | 474 | 227 | 136 | 923 | 602
Participants | 620 | 325 | 169 | 88 | 685 | 428

ADVERSE EVENTS:
Description: Study was divided into Part A and Part B and two age strata, 50-64 and 65 and older. Only subjects that completed Part A were allowed to enroll in Part B. Per SAP the analyses were performed by treatment group and age stratum, in addition it was pre-determined to also present AEs for those subjects that received both the VCIV + EIV per age stratum.
Arm/Group | VCIV (50-64 Years) | VCIV (65+ Years) | EIV (50-64 Years) | EIV (65+ Years) | VCIV + EIV (50-64 Years) | VCIV + EIV (65+ Years)
All-Cause Mortality (participants affected / at risk) | 1/828 | 3/474 | 0/227 | 0/136 | 1/923 | 1/602
Serious Adverse Events (participants affected / at risk) | 32/828 | 28/474 | 4/227 | 10/136 | 25/923 | 32/602
Other Adverse Events (participants affected / at risk) | 777/828 | 297/474 | 183/227 | 95/136 | 492/923 | 346/602
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VCIV (50-64 Years) (N=828) | VCIV (65+ Years) (N=474) | EIV (50-64 Years) (N=227) | EIV (65+ Years) (N=136) | VCIV + EIV (50-64 Years) (N=923) | VCIV + EIV (65+ Years) (N=602)
Electromechanical dissociation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 2 | 0 | 2 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abscess rupture (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0 | 0 | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back injury (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 3
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2
Chest pain (Cardiac disorders) | 1 | 1 | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colon neoplasm (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Implantable defibrillator malfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 3
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Rectal polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haematoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sick sinus syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Surgical failure (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thyroid adenoma (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Transient ischaemic attack (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VCIV (50-64 Years) (N=828) | VCIV (65+ Years) (N=474) | EIV (50-64 Years) (N=227) | EIV (65+ Years) (N=136) | VCIV + EIV (50-64 Years) (N=923) | VCIV + EIV (65+ Years) (N=602)
Cough (Respiratory, thoracic and mediastinal disorders) | 123 | 46 | 16 | 13 | 60 | 44
Diarrhea (Gastrointestinal disorders) | 72 | 39 | 13 | 4 | 37 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 209 | 81 | 27 | 8 | 14 | 11
Chills (General disorders) | 217 | 86 | 21 | 6 | 17 | 5
Fatigue (General disorders) | 448 | 178 | 53 | 19 | 14 | 9
Headache (Nervous system disorders) | 510 | 166 | 70 | 18 | 73 | 31
Hyperhidrosis (Nervous system disorders) | 164 | 43 | 14 | 4 | 2 | 0
Hypertension (Vascular disorders) | 60 | 53 | 12 | 10 | 15 | 15
Injection site pain (General disorders) | 560 | 173 | 69 | 30 | 36 | 14
Malaise (General disorders) | 451 | 176 | 48 | 16 | 9 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 369 | 138 | 48 | 12 | 17 | 9
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 64 | 35 | 17 | 11 | 56 | 27
Nausea (Gastrointestinal disorders) | 71 | 34 | 9 | 1 | 36 | 14
Oropharyngeal pain (Nervous system disorders) | 128 | 48 | 16 | 15 | 61 | 25
Pyrexia (General disorders) | 91 | 36 | 16 | 3 | 33 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 59 | 35 | 15 | 7 | 48 | 31
Upper respiratory tract infection (Infections and infestations) | 74 | 47 | 31 | 11 | 62 | 47
Blood pressure increased (Vascular disorders) | 73 | 30 | 8 | 5 | 5 | 9
Injection site erythema (General disorders) | 70 | 38 | 6 | 5 | 10 | 1
Injection site swelling (General disorders) | 77 | 40 | 5 | 3 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 80 | 20 | 11 | 7 | 12 | 30
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 47 | 14 | 8 | 9 | 43 | 14
Vomiting (Gastrointestinal disorders) | 59 | 31 | 8 | 1 | 30 | 143
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 19 | 8 | 23 | 7 | 15
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 24 | 16 | 10 | 6 | 21 | 22
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 51 | 20 | 6 | 1 | 26 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes